CLINICAL TRIAL: NCT02801539
Title: Respiratory Muscle Training in Late-Onset Pompe Disease
Brief Title: Respiratory Muscle Training in L-Onset Pompe Disease (LOPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00068728; 1R21AR069880-01 (NIH)
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Glycogen Storage Disease Type II
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory muscle training (RMT) (Experimental): Subjects in the experimental arm will be given an inspiratory and expiratory RMT device to use during Duke-based and home-based RMT therapy.
  Interventions: Device: RMT therapy using modified RMT device
- Sham-RMT (Sham Comparator): Subjects in control arm will be given an inspiratory and expiratory sham-device and will complete Duke-based and home-based sham-RMT therapy.
  Interventions: Device: Sham-RMT therapy using modified RMT device

INTERVENTIONS:
Device: RMT therapy using modified RMT device — The exercises provided by the RMT device is intended to strengthen breathing muscles.
  Arms: Respiratory muscle training (RMT)
Device: Sham-RMT therapy using modified RMT device — The exercises provided by the Sham-RMT modified device is not intended to strengthen breathing muscles.
  Arms: Sham-RMT

SUMMARY:
This study is being done to test the effects of respiratory muscle training (RMT) in patients with late-onset Pompe Disease (LOPD) who have weakness of their breathing muscles. The results of this study will help design future research studies about RMT in LOPD. The goals of this study are to decide if sham-RMT is a useful control condition for RMT and to choose the best ways to measure the health benefits of RMT in LOPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of LOPD
* On enzyme replacement therapy for ≥ 26 weeks at pretest
* Able to follow directions for study participation
* Able to complete a home-based RMT regimen

Exclusion Criteria:

* Neurodegenerative conditions (e.g. stroke, dementia) or other serious neurologic condition that would prevent meaningful study participation as determined at the discretion of the principle investigator
* Inability to give legally effective consent
* Inability to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Change in respiratory strength | baseline, 12 weeks, 6 months, 9 months
  RMT to sham-RMT comparison of maximum inspiratory pressures (MIP). Change pretest to posttest is primary measure (baseline to 12 weeks).
Feasibility of sham-RMT, as measured by program adherence | 12 weeks
  As measured by program adherence (good is considered greater than or equal to 80%). Helps determines if a future efficacy trial is warranted and if sham-RMT may be a good control condition for a future trial.

SECONDARY OUTCOMES:
Change in maximum expiratory pressures (MEP) | baseline, 12 weeks, 6 months, 9 months
  Change pretest to posttest
Change in 6-minute walk test (6MWT) | baseline, 12 weeks, 6 months, 9 months
  Change pretest to posttest
Change in Gait, Stairs, Gower, and Chair (GSGC) scale | baseline, 12 weeks, 6 months, 9 months
  Change pretest to posttest
Change in peak cough flow (PCF) | baseline, 12 weeks, 6 months, 9 months
  Change pretest to posttest
Change in Rasch-built Pompe-specific Activity Score (R-PAct) | baseline, 12 weeks, 6 months, 9 months
  Change pretest to posttest
Change in diaphragm thickness | baseline, 12 weeks, 6 months, 9 months
  change pretest to posttest

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Jones, PhD, Principal Investigator — Division of Head and Neck Surgery & Communication Sciences, Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones HN, Kuchibhatla M, Crisp KD, Hobson Webb LD, Case L, Batten MT, Marcus JA, Kravitz RM, Kishnani PS. Respiratory muscle training (RMT) in late-onset Pompe disease (LOPD): A protocol for a sham-controlled clinical trial. Mol Genet Metab. 2019 Aug;127(4):346-354. doi: 10.1016/j.ymgme.2019.05.001. Epub 2019 May 8. PMID 31303277